CLINICAL TRIAL: NCT03271398
Title: Intensive Therapy Archival Research
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trauma Institute & Child Trauma Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 2017-1001
Record Dates: First submitted 2017-08-31; First posted 2017-09-05 (Actual); Last update posted 2017-09-07 (Actual); Status verified 2017-09

CONDITIONS: Trauma, Psychological
MeSH Terms: conditions — Psychological Trauma | interventions — Eye Movement Desensitization Reprocessing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Adult victims of sexual assault
  Interventions: Behavioral: EMDR; Behavioral: PC
- Children who have been exposed to domestic abuse
  Interventions: Behavioral: EMDR; Behavioral: PC
- Women with perinatal emotional complications
  Interventions: Behavioral: EMDR; Behavioral: PC
- Teens with behavior problems and histories of abuse
  Interventions: Behavioral: EMDR; Behavioral: PC
- Veterans with military-related trauma
  Interventions: Behavioral: EMDR; Behavioral: PC
- Survivors of intimate partner violence
  Interventions: Behavioral: EMDR; Behavioral: PC

INTERVENTIONS:
Behavioral: EMDR — Eye movement desensitization and reprocessing (intensive format)
Behavioral: PC — Progressive counting (intensive format)

SUMMARY:
This is an internal treatment evaluation to determine whether eye movement desensitization and reprocessing (EMDR) or progressive counting (PC) should become the preferred trauma treatment for the investigator's clients. The investigator is using routine/existing in-house measures and case files to track symptom reduction, trauma treatment time, rate of treatment switching (from EMDR to PC or vice versa), and rate of trauma treatment refusal. This is retrospective as well as prospective archival research.

ELIGIBILITY:
Inclusion Criteria:

* Victims of crimes, including assault, rape, robbery, intimate partner violence, child abuse, kidnapping, vehicular homicide, and suicide
* Witnesses and family members of victims

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All participants in the Trauma Institute & Child Trauma Institute Victims of Crime program will be included.
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2017-08-02 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in TSI-2 following treatment | Administered pre-treatment, two weeks post-treatment, and 12 weeks post-treatment
  Trauma Symptom Inventory-2
Change in TSCC following treatment | Administered pre-treatment, two weeks post-treatment, and 12 weeks post-treatment
  Trauma Symptom Checklist for Children
Change in PRS following treatment | Administered pre-treatment, two weeks post-treatment, and 12 weeks post-treatment
  Problem Rating Scale

CONTACTS AND LOCATIONS:
Overall Officials: Ricky Greenwald, PsyD, Principal Investigator — Trauma Institute & Child Trauma Institute
Locations (1):
- Trauma Institute & Child Trauma Institute, Northampton, Massachusetts, United States

REFERENCES:
- [Derived] Greenwald R, Camden AA. A pragmatic randomized comparison of intensive EMDR and intensive PC for victims of crime. Psychol Trauma. 2024 Jan;16(1):134-142. doi: 10.1037/tra0001176. Epub 2022 Feb 10. PMID 35143219